CLINICAL TRIAL: NCT04890509
Title: A Multicentre, Phase 2, Randomised Study to Assess the Efficacy and Safety of Bemcentinib for the Treatment of COVID-19 in Hospitalised Patients
Brief Title: A Study of Bemcentinib for the Treatment of COVID-19 in Hospitalised Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BerGenBio ASA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGBC020
Record Dates: First submitted 2021-05-17; First posted 2021-05-18 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — bemcentinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care + Bemcentinib (Experimental): Bemcentinib will be administered for up to 15 days, or until discharge from hospital, whichever comes sooner. SoC will be administered based on local guidelines.
  Interventions: Drug: Bemcentinib; Other: SoC
- Standard of Care (Active Comparator): The SoC will be administered based on local guidelines in place at the time of treatment during the study.
  Interventions: Other: SoC

INTERVENTIONS:
Drug: Bemcentinib — Bemcentinib capsules will be administered orally.
  Arms: Standard of Care + Bemcentinib
Other: SoC — The SoC will be administered based on local guidelines.

SUMMARY:
The primary objective of the study is to evaluate the efficacy of bemcentinib as an add-on therapies to standard of care (SoC) in participants hospitalized with coronavirus disease 2019 (COVID-19).

ELIGIBILITY:
Inclusion Criteria:

* Adults (greater than or equal to [>=] 18 years) with SARS-CoV-2 infection.
* Participants with symptoms and/or signs consistent with COVID-19, requiring treatment.
* A score of Grade 3 to 5 on the 9-point ordinal scale. In India; only Participants with a score of Grade 4 or 5 will be enrolled.
* a) Male Participants:
* A male Participant must agree to use contraception during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.

  b) Female Participants:
* A female Participant is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

  1. Not a woman of childbearing potential. OR
  2. A woman of childbearing potential who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment.
* Women who are lactating who agree not to breastfeed their child during the study and for at least 120 days after termination of study therapy (they may continue to express milk away from the child during this period, but this milk must be discarded).
* Ability to provide informed consent signed by the study Participant or legally authorized representative.

Exclusion Criteria:

* Participants who have previously had a score of 6 or 7 on the 9-point ordinal scale.
* Inability to swallow capsules (administration via nasogastric tube is permitted in Participants who become unable to swallow after starting the study drug).
* History of the following cardiac conditions:

  1. Myocardial infarction within 3 months prior to the first dose
  2. Unstable angina
  3. History of clinically significant dysrhythmias (long QT features on electrocardiogram [ECG], sustained bradycardia [less than or equal to {<=} 55 beats per minute {bpm}]), left bundle branch block, or ventricular arrhythmia) or history of familial long QT. Participants with an implantable cardioverter defibrillator device in place, will be allowed to enroll. Atrial fibrillation will not be a reason for exclusion.
* Screening 12-lead ECG with a measurable QT interval according to Fridericia correction (QTcF) greater than (>) 470 msec.
* Clinically significant hypokalaemia.
* Therapeutic anticoagulation with vitamin K antagonists.
* Previous bowel resection that would interfere with drug absorption.
* Any participant whose interests are not best served by study participation, as determined by a senior attending clinician.
* Alanine aminotransferase/aspartate aminotransferase >5 × the upper limit of normal.
* Current treatment for human immunodeficiency virus (HIV) or tuberculosis (TB).
* Positive serologic assay at screening for hepatitis B virus (Hep B surface antigen) or hepatitis C virus (hepatitis C PCR or hepatitis C core antigen) at local laboratory.
* Stage 4 severe chronic kidney disease.
* Anticipated transfer to another hospital that is not a study center within 72 hours.
* Allergy to any study treatment.
* Experimental off-label usage of medicinal products as treatments for COVID-19 at the time of enrolment.
* Participants participating in another clinical study of an investigational medicinal product.
* Current or planned treatment for TB.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hani Gabra, Study Chair — BerGenBio ASA
Locations (12):
- India (7):
  - Unity Trauma Center and ICU, Unity Hospital, Surat, Gujarat
  - Kasturba Medical College, Mangalore, Karnataka
  - JSS Hospital, Mysuru, Karnataka
  - Chopda Medicare & Research Centre Pvt. Ltd (CMARC) - Magnum Heart Institute, Nashik, Maharashtra
  - Sahyadri Specialty Hospital, Pune, Maharashtra
  - Krishna Institute of Medical Sciences (KIMS Hospitals), Secunderabad, Telangana
  - Maulana Azad Medical College, New Delhi
- South Africa (5):
  - Lakeview Hospital, Mowbray, Benoni
  - Tiervlei Trial Centre, Bellville, Cape Town
  - Vergelegen Mediclinic, Somerset West, Cape Town
  - Into Research, Groenkloof, Pretoria
  - Clinical Projects Research, Worcester

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification [text, tables, figures and appendices].
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Proposal should be directed to HYPERLINK "mailto:clinical@bergenbio.com" clinical@bergenbio.com. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Groups:
- Bemcentinib + Standard of Care (SoC): Bemcentinib was administered for up to 15 days, or until discharge from hospital, whichever came sooner. SoC was administered based on local guidelines.
- Standard of Care: The SoC was administered based on local guidelines in place at the time of treatment during the study.
Period: Overall Study
Arm/Group | Bemcentinib + Standard of Care (SoC) | Standard of Care
Started | 58 | 57
Completed | 54 | 53
Not Completed | 4 | 4
Not completed — Death | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bemcentinib + Standard of Care (SoC) | Standard of Care | Total
Number analyzed (Participants) | 58 | 57 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (12.97) | 51.5 (15.48) | 53.0 (14.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 22 | 39
  Male | 41 | 35 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 57 | 56 | 113
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Time to Sustained Clinical Improvement of at Least 2 Points
Description: Sustained clinical improvement is defined as improvement without subsequent worsening. Time to sustained clinical improvement (in days) from randomization is defined as the number of days to a sustained improvement of at least 2 points on a 9-point category ordinal scale, or live discharge from the hospital, or fit for discharge, whichever occurs first by Day 29. 9-point category ordinal scale: 0-Uninfected, no clinical or virological evidence of infection; 1-Ambulatory, no limitation of activities; 2-Ambulatory, limitation of activities; 3-Hospitalised - mild disease, no oxygen therapy; 4-Hospitalized - mild disease, oxygen by mask or nasal prongs; 5-Hospitalized - severe disease, non-invasive ventilation or high-flow oxygen; 6-Hospitalized - severe disease, intubation and mechanical ventilation; 7-Hospitalized - severe disease, ventilation and additional organ support - vasopressors, renal replacement therapy, extracorporeal membrane oxygenation; 8-Death.
Time Frame: From randomization up to Day 29
Population: Intention to treat (ITT) analysis set included all participants who were randomized and matched the inclusion/exclusion criteria of the protocol. Here, 'N' (overall number of participants analyzed) is defined as participants who were evaluable for this outcome measure.
Measure: Median (80% Confidence Interval); unit: days
Arm/Group | Bemcentinib + Standard of Care (SoC) | Standard of Care
Number analyzed (Participants) | 54 | 53
days | 7.0 [6.00 to 8.00] | 7.0 [6.00 to 9.00]

2. Secondary Outcome: Percentage of Participants Not Deteriorating According to the Ordinal Scale by 1, 2, or 3 Points
Description: Percentage of participants not deteriorating according to the 9-point category Ordinal Scale (0= uninfected and 8= Death), by 1, 2, or 3 points was reported. Deterioration by 1, 2 or 3 points at days 2, 8, 15 and 29 is defined as an increase in ordinal scale score of at least 1, 2 or 3 points respectively compared to baseline. Participants who had no ordinal score measured at a Day and who were discharged from hospital prior to that Day had their ordinal score used from the most recent value recorded prior to the Day. Participants who died prior to a Day have a score of 8 used for all Days after death. All other participants with no ordinal score measured at a day are considered to have deterioration at that Day.
Time Frame: At Days 2, 8, 15, and 29
Population: Population included ITT analysis set.
Measure: Number; unit: Percentage of participants
Arm/Group | Bemcentinib + Standard of Care (SoC) | Standard of Care
Number analyzed (Participants) | 58 | 57
Percentage of participants
  Day 2: deterioration of 1 point | 95.7 | 86.0
  Day 8: deterioration of 1 point | 96.6 | 87.7
  Day 15: deterioration of 1 point | 96.6 | 91.2
  Day 29: deterioration of 1 point | 94.8 | 94.7
  Day 2: deterioration of 2 point | 99.3 | 100.0
  Day 8: deterioration of 2 point | 100.0 | 93.0
  Day 15: deterioration of 2 point | 98.3 | 93.0
  Day 29: deterioration of 2 point | 94.8 | 94.7
  Day 2: deterioration of 3 point | 99.5 | 100.0
  Day 8: deterioration of 3 point | 100.0 | 96.5
  Day 15: deterioration of 3 point | 100.0 | 94.7
  Day 29: deterioration of 3 point | 96.6 | 94.7

3. Secondary Outcome: Duration of Oxygen Use (in Percentage)
Description: In this outcome measure percentage of hospitalization days during which oxygen was used is reported. The duration of each occurrence of oxygen use was derived based on the start date and time, and end date and time of the use of any type of supplemental oxygen (including mechanical ventilation) as captured in the electronic case report form (eCRF). For each participant, the duration in days of oxygen use was derived as the sum of the duration (in minutes) of each occurrence of oxygen use, divided by 1440 (24*60).
Time Frame: Up to Day 29
Population: Population included ITT analysis set.
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Bemcentinib + Standard of Care (SoC) | Standard of Care
Number analyzed (Participants) | 58 | 57
Percentage of days | 53.33 (30.572) | 56.38 (30.641)

4. Secondary Outcome: Duration of Oxygen-free Days (in Percentage)
Description: In this outcome measure percentage of hospitalization days which were oxygen-free days was reported.
Time Frame: Up to Day 29
Population: Population included ITT analysis set.
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Bemcentinib + Standard of Care (SoC) | Standard of Care
Number analyzed (Participants) | 58 | 57
Percentage of days | 46.67 (30.572) | 43.62 (30.641)

5. Secondary Outcome: Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Viral Load
Description: SARS-CoV-2 viral load was determined by polymerase chain reaction (PCR) in oropharyngeal and nasal swab while hospitalized. Baseline is defined as the non-missing measurement taken prior to or on randomization day (including unscheduled measurements, if any).
Time Frame: Day 1 (Baseline), 3, 5, 8, 11, 15, and 29
Population: Population included ITT analysis set. Here, 'N' (overall number of participants analyzed) is defined as participants who were evaluable for this outcome measure and 'n' (number analyzed) is defined as number of participants who were analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: copies/milliliter (mL)
Arm/Group | Bemcentinib + Standard of Care (SoC) | Standard of Care
Number analyzed (Participants) | 56 | 54
copies/milliliter (mL)
  Baseline: Oropharyngeal Swab: number analyzed (Participants) | 54 | 53
  Baseline: Oropharyngeal Swab | 18739475 (95276993) | 882663 (3256156)
  Day 3: Oropharyngeal Swab: number analyzed (Participants) | 53 | 50
  Day 3: Oropharyngeal Swab | 2293266 (15729688) | 5081599 (25118620)
  Day 5: Oropharyngeal Swab: number analyzed (Participants) | 39 | 29
  Day 5: Oropharyngeal Swab | 140383 (666211) | 742869 (3152847)
  Day 8: Oropharyngeal Swab: number analyzed (Participants) | 36 | 27
  Day 8: Oropharyngeal Swab | 13897399 (83331884) | 7021884 (35625407)
  Day 11: Oropharyngeal Swab: number analyzed (Participants) | 15 | 19
  Day 11: Oropharyngeal Swab | 53745 (192226) | 1304145 (3812646)
  Day 15: Oropharyngeal Swab: number analyzed (Participants) | 37 | 23
  Day 15: Oropharyngeal Swab | 15124 (58315) | 31707 (136984)
  Day 29: Oropharyngeal Swab: number analyzed (Participants) | 39 | 35
  Day 29: Oropharyngeal Swab | 500 (0) | 154574 (884358)
  Baseline: Nasopharyngeal Swab | 7374030 (35266724) | 18685634 (82429609)
  Day 3: Nasopharyngeal Swab: number analyzed (Participants) | 54 | 51
  Day 3: Nasopharyngeal Swab | 1073239 (4768036) | 13012043 (71173469)
  Day 5: Nasopharyngeal Swab: number analyzed (Participants) | 40 | 31
  Day 5: Nasopharyngeal Swab | 7161257 (33851537) | 18143671 (89821021)
  Day 8: Nasopharyngeal Swab: number analyzed (Participants) | 36 | 28
  Day 8: Nasopharyngeal Swab | 435108 (1581546) | 987743 (4274477)
  Day 11: Nasopharyngeal Swab: number analyzed (Participants) | 14 | 18
  Day 11: Nasopharyngeal Swab | 160017 (579053) | 434152 (1797045)
  Day 15: Nasopharyngeal Swab: number analyzed (Participants) | 34 | 24
  Day 15: Nasopharyngeal Swab | 28730 (117210) | 10974 (24096)
  Day 29: Nasopharyngeal Swab: number analyzed (Participants) | 37 | 33
  Day 29: Nasopharyngeal Swab | 995 (1389) | 1218 (3170)

6. Secondary Outcome: Duration of Ventilation Use (in Percentage) by Hospital Survival Status
Description: In this outcome measure percentage of hospitalization days during which ventilation was used. Duration of ventilation use by hospital survival status was reported in terms of days. Alive is defined as a participant who did not die whilst in hospital and died is defined as a participant who died whilst in hospital. The duration of ventilation was derived based on the start date and time, and end date and time of either invasive mechanical ventilation or non-invasive mechanical ventilation as the type of supplemental oxygen captured in the eCRF.
Time Frame: Up to Day 29
Population: Population included ITT analysis set. Here, 'n' (number analyzed) is defined as number of participants who were analyzed for specified category per hospital survival status.
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Bemcentinib + Standard of Care (SoC) | Standard of Care
Number analyzed (Participants) | 58 | 57
Percentage of days
  Alive: number analyzed (Participants) | 56 | 53
  Alive | 1.68 (12.592) | 6.20 (18.952)
  Died: number analyzed (Participants) | 2 | 4
  Died | 31.36 (44.353) | 73.99 (19.652)

7. Secondary Outcome: Duration of Ventilation-free Days (in Percentage)- by Hospital Survival Status
Description: In this outcome measure percentage of hospitalization days which were ventilation-free by hospital survival status was reported. Alive is defined as a participant who did not die whilst in hospital and died is defined as a participant who died whilst in hospital.
Time Frame: Up to Day 29
Population: Population included ITT analysis set. Here, 'n' (number analyzed) is defined as number of participants who were analyzed in specified category per hospital survival status.
Measure: Median (Standard Deviation); unit: Percentage of days
Arm/Group | Bemcentinib + Standard of Care (SoC) | Standard of Care
Number analyzed (Participants) | 58 | 57
Percentage of days
  Alive: number analyzed (Participants) | 56 | 53
  Alive | 98.32 (12.592) | 93.80 (18.952)
  Died: number analyzed (Participants) | 2 | 4
  Died | 68.64 (44.353) | 26.01 (19.652)

8. Secondary Outcome: Number of Participants With Any Form of New Ventilation Use
Description: Number of participants with any form of new ventilation use was reported. New ventilation was defined as either Invasive Mechanical Ventilation or Non-Invasive Mechanical Ventilation as the type of supplemental oxygen captured in the eCRF that was not occurring at the time of randomization.
Time Frame: Up to Day 29
Population: Population included ITT analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Bemcentinib + Standard of Care (SoC) | Standard of Care
Number analyzed (Participants) | 58 | 57
Participants | 1 | 6

9. Secondary Outcome: Duration of New Ventilation Use (in Percentage) by Hospital Survival Status
Description: In this outcome measure percentage of hospitalization days during which new ventilation was used. The duration of new ventilation was derived based on the start date and time, and end date and time of either invasive mechanical ventilation or non-invasive mechanical ventilation as the type of supplemental oxygen captured in the eCRF that was not occurring at the time of randomization. Alive is defined as a participant who did not die whilst in hospital and died is defined as a participant who died whilst in hospital.
Time Frame: Up to Day 29
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Bemcentinib + Standard of Care (SoC) | Standard of Care
Number analyzed (Participants) | 58 | 57
Percentage of days
  Alive: number analyzed (Participants) | 56 | 53
  Alive | 0.00 (0.000) | 3.26 (13.666)
  Died: number analyzed (Participants) | 2 | 4
  Died | 31.36 (44.353) | 46.96 (35.463)

10. Secondary Outcome: Duration of Organ Support (in Percentage)
Description: In this outcome measure percentage of hospitalization days during which organ support (e.g., including respiratory, renal, and cardiac support) was provided is reported in days. Organ support was approximated from the following adverse events of special interests (AESIs) when treatment was received: Cardiovascular organ failure; Renal organ failure requiring renal replacement therapy; Liver organ failure. For each participant the duration of AESIs was summed, noting that if there are any overlapping dates of AESIs, days were only counted once for a participant.
Time Frame: Up to Day 29
Population: Population included ITT analysis set.
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Bemcentinib + Standard of Care (SoC) | Standard of Care
Number analyzed (Participants) | 58 | 57
Percentage of days | 1.0 (4.73) | 1.0 (3.19)

11. Secondary Outcome: Number of Participants With Response
Description: Response rate was assessed on a 9-point category ordinal scale. Number of participants with response (defined as sustained clinical improvement of at least 2 points (from randomization) on a 9-point category ordinal scale, live discharge from the hospital, or considered fit for discharge (a score of 0, 1, or 2 on the ordinal scale), whichever comes first) was reported. Participants who were not discharged or who had no ordinal scale assessment on a particular study day (including participants who have died prior to that study day) were considered non-responders.
Time Frame: At Days 2, 8, 15, and 29
Population: Population included ITT analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Bemcentinib + Standard of Care (SoC) | Standard of Care
Number analyzed (Participants) | 58 | 57
Participants
  Day 2 | 1 | 4
  Day 8 | 37 | 32
  Day 15 | 54 | 50
  Day 29 | 54 | 53

12. Secondary Outcome: Time to Live Discharge From the Hospital
Description: Time to live discharge from the hospital (in days) was calculated from randomization. It was derived as: (date of discharge - date of randomization) +1. Participants who were alive and still in hospital at the time of analysis had their time to discharge censored at the data cut-off date for the analysis. Participants who died at the time of analysis, without having been discharged from hospital, had their time to live discharge censored at Day 29.
Time Frame: Up to Day 29
Population: Population included ITT analysis set.
Measure: Median (80% Confidence Interval); unit: days
Arm/Group | Bemcentinib + Standard of Care (SoC) | Standard of Care
Number analyzed (Participants) | 58 | 57
days | 7.0 [6.00 to 8.00] | 7.0 [6.00 to 9.00]

13. Secondary Outcome: Time to Death
Description: Time to death (in days) was calculated from randomization. Participants who were not known to have died at the time of analysis had their time to death censored at the last date the participant was known to be alive.
Time Frame: Up to Day 60
Population: Population included ITT analysis set.
Measure: Median (80% Confidence Interval); unit: days
Arm/Group | Bemcentinib + Standard of Care (SoC) | Standard of Care
Number analyzed (Participants) | 58 | 57
days | NA [NA to NA] — Here, NA signifies that median and confidence interval (CI) was not estimable due to fewer number of events. | NA [NA to NA] — Here, NA signifies that median and confidence interval (CI) was not estimable due to fewer number of events.

14. Secondary Outcome: Overall Mortality
Description: Number of participants who died were reported.
Time Frame: At Days 15, 29, and 60
Population: Population included ITT analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Bemcentinib + Standard of Care (SoC) | Standard of Care
Number analyzed (Participants) | 58 | 57
Participants
  Day 15 | 1 | 3
  Day 29 | 2 | 3
  Day 60 | 4 | 4

15. Secondary Outcome: Change From Baseline in the Ratio of Oxygen Saturation to Fraction of Inspired Oxygen Concentration (SpO2/FiO2)
Description: Change from baseline in the ratio of the oxygen saturation to fraction of inspired oxygen concentration (SpO2/FiO2) was measured daily from randomization to Day 15. Baseline is defined as the last non-missing measurement taken prior to randomization (including unscheduled measurements, if any).
Time Frame: Baseline, Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: Population included ITT analysis set. Here, 'N' (overall number of participants analyzed) is defined as participants who were evaluable for this outcome measure and 'n' (number analyzed) is defined as number of participants analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Bemcentinib + Standard of Care (SoC) | Standard of Care
Number analyzed (Participants) | 25 | 28
ratio
  Day 2: number analyzed (Participants) | 25 | 26
  Day 2 | 1.65 (6.697) | -6.21 (28.529)
  Day 3: number analyzed (Participants) | 22 | 28
  Day 3 | 2.31 (10.623) | -2.57 (51.482)
  Day 4: number analyzed (Participants) | 25 | 23
  Day 4 | 2.82 (49.619) | -23.03 (72.541)
  Day 5: number analyzed (Participants) | 21 | 22
  Day 5 | -44.45 (91.184) | -35.72 (107.087)
  Day 6: number analyzed (Participants) | 14 | 21
  Day 6 | -107.54 (103.717) | -42.52 (119.974)
  Day 7: number analyzed (Participants) | 16 | 20
  Day 7 | -93.13 (129.911) | -50.60 (127.830)
  Day 8: number analyzed (Participants) | 14 | 18
  Day 8 | -118.03 (107.490) | -67.97 (113.665)
  Day 9: number analyzed (Participants) | 16 | 15
  Day 9 | -99.87 (114.115) | -79.17 (126.275)
  Day 10: number analyzed (Participants) | 11 | 14
  Day 10 | -143.88 (111.903) | -83.25 (129.137)
  Day 11: number analyzed (Participants) | 12 | 14
  Day 11 | -130.46 (94.651) | -90.87 (121.258)
  Day 12: number analyzed (Participants) | 11 | 12
  Day 12 | -116.99 (118.048) | -99.57 (129.758)
  Day 13: number analyzed (Participants) | 6 | 6
  Day 13 | -145.17 (127.030) | -132.79 (100.626)
  Day 14: number analyzed (Participants) | 3 | 4
  Day 14 | -196.58 (5.627) | -120.55 (138.842)
  Day 15: number analyzed (Participants) | 6 | 6
  Day 15 | -109.43 (203.712) | -109.35 (134.538)

16. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in participants, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: Up to Day 90
Population: Safety analysis set included all participants who were randomized and received at least 1 dose of study treatment (bemcentinib or SoC).
Measure: Count of Participants; unit: Participants
Arm/Group | Bemcentinib + Standard of Care (SoC) | Standard of Care
Number analyzed (Participants) | 58 | 57
Participants | 18 | 22

17. Secondary Outcome: Duration of Intensive Care Unit (ICU)- (in Percentage)
Description: In this outcome measure percentage of hospitalization days for which participant was in ICU is reported. Duration of ICU was derived based on start/stop date of admission and start/stop date of ICU stay in the eCRF. Duration of ICU is the sum of duration (days) of each episode of ICU/HDU stay. If a participant died and the stop date of admission is missing, the date of death was used instead.
Time Frame: Up to 90 days
Population: Population included ITT analysis set.
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Bemcentinib + Standard of Care (SoC) | Standard of Care
Number analyzed (Participants) | 58 | 57
Percentage of days | 32.03 (44.234) | 40.89 (45.668)

18. Secondary Outcome: Duration of Hospitalization
Description: Duration of hospitalization (days) was derived based on start/stop date of admission and start/stop date of HDU stay in the eCRF. Duration of hospitalization is derived as stop date of admission minus start date of admission +1. If a participant died and the stop date of admission is missing, the date of death was used instead.
Time Frame: Up to 90 days
Population: Population included ITT analysis set.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bemcentinib + Standard of Care (SoC) | Standard of Care
Number analyzed (Participants) | 58 | 57
days | 9.8 (5.68) | 10.5 (5.77)

19. Secondary Outcome: National Early Warning Score 2 (NEWS2)
Description: NEWS2 is based on 6 physiological measurements (respiration rate, oxygen saturation [SpO2], systolic blood pressure, pulse rate, level of consciousness or new confusion, and temperature). Each of these physiological parameters is rated using a 4-point Likert scale (0= no risk to 3 = high risk). The NEWS2 score is obtained by summing the 6 physiological parameter individual scores, with higher score indicating higher risk of deterioration and need for escalation in clinical care, including transfer of the participant to a higher level of care hospital unit. The NEWS2 score is set to missing if at least 1 physiological parameter individual score is missing, and the overall score is uplifted by 2 points for patients requiring supplemental oxygen to maintain their recommended SpO2. The range of NEWS2 score, taking into account this potential 2 point uplifting, is 0 (best) to 20 (worst).
Time Frame: At Days 15 and 29
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bemcentinib + Standard of Care (SoC) | Standard of Care
Number analyzed (Participants) | 31 | 29
units on a scale
  Day 15: number analyzed (Participants) | 14 | 13
  Day 15 | 1.8 (3.29) | 2.2 (2.62)
  Day 29 | 0.8 (1.50) | 0.7 (1.49)

20. Secondary Outcome: Time to NEWS2 of <=2, Maintained for at Least 24 Hours
Description: The NEWS2 is based on is based on 6 physiological measurements. The range of NEWS2 score, is from 0 (best) to 20 (worst). Time to NEWS2 <=2 maintained for at least 24 hours (in days) was calculated from randomization as: The date of the first post-Baseline assessment where NEWS2 is <= 2 and sustained for at least 24 hours ) - date of randomization +1.
Time Frame: Up to Day 29
Population: Population included ITT analysis set.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Bemcentinib + Standard of Care (SoC) | Standard of Care
Number analyzed (Participants) | 58 | 57
days | 4.0 [4.00 to 5.00] | 4.0 [3.00 to 8.00]

21. Secondary Outcome: Ranked Trajectory Over 29 Days
Description: Ranked trajectory is not a scale outcome measure and does not have a validated scale range. It is an evaluation of dynamic changes over time in the ordinal scale (9-point; 0= uninfected to 8= death; higher scores = more severity) of severity based on individual rank. It was calculated over 29 days. Each participant ranks were assigned based on the following order of the ordinal scale, [1] The worst (highest) score, Ascending; [2] The last recorded score, Ascending; [3] The number of days at worst score, Ascending; [4] The best(lowest) score that occurred after the worst score, Ascending; [5] The number of days the participant was at [4], Descending. Orderings performed at steps [2], [3], [4] and [5] were used to resolve any tied ranks resulting from previous step. Each participant had one overall rank for their trajectory. There was no rank range associated, however lower rank = better trajectory.
Time Frame: 29 days
Population: Population included ITT analysis set.
Measure: Mean (Standard Error); unit: rank score
Arm/Group | Bemcentinib + Standard of Care (SoC) | Standard of Care
Number analyzed (Participants) | 58 | 57
rank score | 58.2 (4.20) | 57.8 (4.66)

ADVERSE EVENTS:
Time Frame: up to Day 90
Description: Safety analysis set included all participants who were randomized and received at least 1 dose of study treatment (bemcentinib or SoC).
Arm/Group | Bemcentinib + Standard of Care (SoC) | Standard of Care
All-Cause Mortality (participants affected / at risk) | 4/58 | 4/57
Serious Adverse Events (participants affected / at risk) | 6/58 | 4/57
Other Adverse Events (participants affected / at risk) | 18/58 | 22/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bemcentinib + Standard of Care (SoC) (N=58) | Standard of Care (N=57)
Cardiac arrest (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Death (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 0 | 2
Aspergillus infection (Infections and infestations) | 1 | 0
Candida infection (Infections and infestations) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ischaemic limb pain (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bemcentinib + Standard of Care (SoC) (N=58) | Standard of Care (N=57)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 3 | 0
Hypercoagulation (Blood and lymphatic system disorders) | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Constipation (Gastrointestinal disorders) | 3 | 1
Anal inflammation (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Impetigo (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Acoustic neuritis (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 3
Hypotension (Vascular disorders) | 1 | 1
Haematoma (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's will not discuss or publish trial results after the trial is completed without seeking prior permission of sponsor.

DOCUMENTS (2):
  • Study Protocol (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/09/NCT04890509/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/09/NCT04890509/SAP_001.pdf